CLINICAL TRIAL: NCT03147105
Title: Armergometry to Improve Mobility in Chronic Progressive Multiple Sclerosis
Brief Title: Armergometry to Improve Mobility in MS
Acronym: AMBOS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Collaborators: Deutsche Multiple Sklerose Gesellschaft Hamburg (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: inims08
Record Dates: First submitted 2017-03-02; First posted 2017-05-10 (Actual); Last update posted 2017-05-30 (Actual); Status verified 2017-05

CONDITIONS: Multiple Sclerosis
Keywords: chronic progressive multiple sclerosis, mobility, arm ergometry, rehabilitation
MeSH Terms: conditions — Multiple Sclerosis; Multiple Sclerosis, Chronic Progressive | interventions — Exercise Test

STUDY DESIGN:
Intervention Model Description: waitlist control
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- arm ergometry (Experimental): Home-based treatment after education in center, training following interval training plan on chip cards for 12 weeks at least 4-5 times/week
  Interventions: Behavioral: arm ergometry
- waiting group (Active Comparator): training after 12 weeks.
  Interventions: Behavioral: arm ergometry

INTERVENTIONS:
Behavioral: arm ergometry — home based arm ergometry, at least 4-5 sessions/week for 12 weeks

SUMMARY:
Chronic progressive multiple sclerosis patients will be randomised to home-based arm ergometry training for 12 weeks or a waitlist control group which will have access to the treatment after 12 weeks when primary endpoint assessment has been obtained. Assessments include clinical outcomes and questionnaires as well MRI imaging and transcranial magnetic stimulation paradigms. Primary endpoint will be the 6 minute walking test at week 12.

DETAILED DESCRIPTION:
Short protocol Design: Patients with progressive MS (PPMS, SPMS) and moderate disability (Expanded Disability Status Scale 4-6.5) will be randomized to home-based arm ergometry or a waitlist control group. Home-based training will be supervised by SD-card documentation, telephone, email and personal contact.

Inclusion criteria: clinically definite MS according to Poser (1983), no progression in the last 6 months before starting, no acute relapse, age 18- 65 years, EDSS 4-6.5, able to perform all arm- and handfunctions in daily life, able to execute a daily Training.

Exclusion criteria: medical contraindications for exercise therapy like cardiovascular or major orthopedic disease, metal parts in body, substantial cognitive deficit, cardiac pacemaker or other electric implants, pregnancy, epilepsy.

Recruitment sample: n=50 Participants for analysis: n= 40 Control group: Intervention available after 3 months Duration: 3 months, data acquisition until 12 months after intervention Hypothesis: Arm ergometry improves walking ability (measured by 6-Minute Walk Test, 6MWT). Secondary endpoints include cognition, fatigue, depression, life quality and blood markers as BDNF.

Primary endpoint: Walking ability is evaluated before and after the training program (12 weeks) using the 6MWT by measuring the total walking distance within six minutes.

Secondary endpoints:

1. Walking abilities: 25FWT, TUG, 5SST, 9HPT, 7-day-accelerometry, MSWS- 12, Walking analysis on Gaitrite tapestry and with kinect camera with different tasks: normal speed, maximal speed, turning around and double tasking
2. EDSS (Expanded Disability status scale)
3. Fitness measures: areobic fitness (peak oxygen consumption VO2), bioimpedance analysis, DIERS-Myoline Muscle Strength Measurement, dynamic hand force measurement, spiroergometry, accelerometry
4. Neuropsychology: Test battery for Attentional Performance (TAP) including alertness, incompatibility and crossmodal integration, Verbal Learning- and Memory- Test (VLMT), Brief International Cognitive Assessment for MS (BICAMS), Symbol- Digit- Modalities Test (SDMT)
5. Questionnaires: HAQUAMS, Fatigue Scale for Motoric and Cognition (FSMC), Beck- Depressions- Inventar (BDI), Frenchay Activity Index (FAI)
6. cMRT
7. Blood: Neurofilament light, BDNF, Analysis with ELISA

Intervention:

Intervention will be a home-based, individual training with 5 -7 training sessions each week. Each individual training is based on the results of the spiroergometry of the participants. These tests will be conducted at the Competence Center for Sports and Exercise Medicine. The training sessions should be in the areobic exercise sector. In this sector intensity should be conducted at a power, which shows lactate values around 1.5 mmol, RER (Respiratory Exchange Ratio) should be around 0.91 and the subjective stress, measured on Borg-Scale, should be about 11. The V02max should be not higher than 65 %.

Before starting the training at home, patients have to come to the center for adaptation to the training machine, the "Motomed". We will test, if the power for the training estimated from stepwise arm ergometry is adeqaute. The patients will recieve an introduction for motomed as well as information on how to handle the chipcards. Patients will get 3 chipcards with one training program on each. The first card contains 10 training sessions. One training range includes 6 minutes active training followed by 2 minute passive rotation by the motomed. Every minute the direction of the crank changes. The frequency should not be higher than 60- 80 U/min. Patients have to repeat one training range (6min load, 2 minute rest) as often as possible. They will recieve one training plan for orientation. After 4 weeks the patients change the chipcard and they start their training with card number 2. Card number 2 includes the same training program as card number 1, but the power increases about 20-30 %. The results of everyday training will be saved automatically on the chipcards. Stored parameters will be heartrate, the power measured in Watt, the length of the training, the number of training ranges, and the frequency on the crank. Furthermore, patients make notes regarding their results and their perceived exertion during the training (measured by Borg-scaling) on a documentation sheet. If the training is too hard, the patients can either train for a shorter time, they can stop the training or they can use the chipcard with the lower power.

Procedure: After basline-examinations (walking ability, fitness, neuropsychology, blood draw, questionnaires, cMRT without contrast medium), instruction on "Motomed" and training at center, patients will be provided with the machines at their homes and start their training for 12 weeks under supervision (Email, telephone, home visit). Follow-up will be performed with the same assessments as at baseline including stepwise ergometry. For the assessments 2-3 appointments at the center are necessary.

ELIGIBILITY:
Inclusion Criteria:

* proven multiple sclerosis
* stable disease
* EDD 4,0-6,5
* being able to perform arm ergometry

Exclusion Criteria:

* relapse situation
* cognitive deficit unable to understand study
* cardivascular disease
* contraindication for MRI

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2017-05-01 (Actual); Primary Completion 2018-07-01 (Estimated); Study Completion 2018-12-31 (Estimated)

PRIMARY OUTCOMES:
6 minute walking test | 6 min.
  maximum distance in 6 minutes

SECONDARY OUTCOMES:
accelerometry | 7 days
  walking speed through 7 days
verbal learning and memory | 30 minutes
  rapid and delayed recall
peak oxygene uptake | 20 minutes
  at step ergometry
brain atrophy | 3 months
  based on percentage brain volume chnage through 3 months
Brain derived neurotrophic factor | 3 months change
  serum levels

CONTACTS AND LOCATIONS:
Overall Officials: Christoph Heesen, Prof., Principal Investigator — Universitätsklinikum Hamburg-Eppendorf
Locations (1):
- Universitätsklinikum Hamburg-Eppendorf, Hamburg, Germany

IPD SHARING:
Plan to Share IPD: Yes
Enclose access to publication

REFERENCES:
- [Derived] Heinrich I, Rosenthal F, Patra S, Schulz KH, Welsch GH, Vettorazzi E, Rosenkranz SC, Stellmann JP, Ramien C, Pottgen J, Gold SM, Heesen C. Arm Ergometry to Improve Mobility in Progressive Multiple Sclerosis (AMBOS)-Results of a Pilot Randomized Controlled Trial. Front Neurol. 2021 Jul 19;12:644533. doi: 10.3389/fneur.2021.644533. eCollection 2021. PMID 34349716